CLINICAL TRIAL: NCT02278068
Title: A First in Human (FIH) Clinical Study to Assess Safety and Performance of Hepatic Sympathetic Denervation for Treatment of Inadequately Controlled Type 2 Diabetic Subjects on Oral Antihyperglycemic Agents.
Brief Title: COMPLEMENT Study- A First in Human Study of Metabolic Neuromodulation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metavention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MV-2014-ANZ-001
Record Dates: First submitted 2014-10-23; First posted 2014-10-29 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Diabetes; Endocrine, Nutritional and Metabolic Diseases (E00-E89)
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Metabolic Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metabolic Neuromodulation System (MNS) (Experimental): Hepatic sympathetic denervation therapy to aid in glycemic control
  Interventions: Device: Metabolic Neuromodulation System (MNS)

INTERVENTIONS:
Device: Metabolic Neuromodulation System (MNS) — Prospective, First-in-Human (FIH), multi-center, non-randomized trial to evaluate the initial safety and performance of hepatic sympathetic denervation to aid in glycemic control.
  Other Names: Hepatic sympathetic denervation

SUMMARY:
The purpose of this research study is to collect information about a new treatment for Type 2 Diabetes Mellitus (T2DM), using a medical device called the Metabolic Neuromodulation System which is intended to help regulate blood glucose levels in patients whose (T2DM) is not well controlled despite treatment with multiple medications. The medical device delivers low-level radiofrequency energy through the wall of the blood vessel to the liver to disrupt the nerves that lead to the liver. Previous research has shown that disrupting these nerves may lead to a lowering of blood sugar levels.

DETAILED DESCRIPTION:
Prospective, First-in-Human (FIH), multi-center, non-randomized trial to evaluate the initial safety and performance of hepatic sympathetic denervation to aid in glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Uncontrolled T2DM, as evidenced by HbA1c levels, on a consistent oral anti-hyperglycemic drug regimen of at least two different drug classes
* Documented status of stable lifestyle modifications

Exclusion Criteria:

* Diagnosed type 1 diabetes mellitus
* History or diagnosis of proliferative retinopathy or advanced autonomic neuropathy
* Estimated glomerular filtration rate (GFR) < 60mL/min/1.73m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-10; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome as assessed by Incidence of serious adverse device effects | 180 day follow-up
  Incidence of serious adverse device effects

SECONDARY OUTCOMES:
Device and Procedural success | intra operative
  Incidence of successful energy delivery, incidence of serious adverse device effects with 24 hours of procedure
Glycemic control | 180 day and 365 day follow-up
  Number of subjects with a decrease in HbA1c, change in plasma glucose based on fasting glucose and oral glucose tolerance test
Laboratory Assessments/Cardiometabolic Changes | 180 day follow up
  Assessment of chemistry/serum lab values to evaluate safety and performance
Adverse Event Rate | 365 day follow up
  Summary of all reported adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: Mark Webster, Prof, Principal Investigator — Auckland City Hospital
Locations (6):
- New Zealand (6):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Wellington Hospital, Wellington